CLINICAL TRIAL: NCT05645653
Title: Nurse-led Medication Self-management Intervention in the Improvement of Medication Adherence in Adult Patients With Multi-morbidity: A Feasibility Randomized Control Trial
Brief Title: Nurse-led Medication Self-management Intervention in the Improvement of Medication Adherence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hamad Medical Corporation (Industry)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Principal Investigator, Dr. Kalpana Singh, Senior epidemiologist, Hamad Medical Corporation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 296
Record Dates: First submitted 2022-11-20; First posted 2022-12-09 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Heart Diseases; CKD; Diabetes; Cancer; Asthma; Thyroid; Hypertension
MeSH Terms: conditions — Heart Diseases; Diabetes Mellitus; Neoplasms; Asthma; Thyroid Diseases; Hypertension

STUDY DESIGN:
Intervention Model Description: This is a single Centre open label, two-arm randomized controlled trial with 1:1 randomization at the participant level. The patient population will be patients with at least two comorbidities. The patient recruitment will be done in the National Centre for Cancer Care and Research (NCCCR) in the outpatient department in the clinical nurse specialist counselling room.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational treatment (Experimental): The medication self-management intervention consists of three face-to-face education sessions and two weekly telephone follow-up over 6 weeks. Intervention components are derived from an extensive review of the literature, including the related theoretical framework and current practice. Based on the extended IMB model of medication adherence, this intervention is designed to offer information related to medication treatment, motivate patients to adhere, help build medication self-management skills, and develop adherence improvement plans. The face-to-face meeting will take place in the clinical nurse specialist counselling room in NCCCR.
  Interventions: Behavioral: Motivational tteaching
- Standard Care (No Intervention): Participants in the control group will continue to receive standard care from Physicians, nurses, and clinical pharmacists in the NCCCR. Physicians are the primary providers and coordinators of care for patients with chronic conditions. Physicians provide patients consultations and education regarding their diseases and treatments (typically clinician-centred) at each patient visit to the chronic disease clinic.

INTERVENTIONS:
Behavioral: Motivational tteaching — A comprehensive assessment of adherence problems will be firstly conducted to identify the factors that affect adherence, including how and why these factors contribute to poor adherence. Medication-related knowledge and skills will be provided based on individual treatments and barriers to adherence. Motivational interviewing techniques will be used for a better understanding of patients' cognitive factors of adherence behavior.
  Arms: Educational treatment

SUMMARY:
Back ground & Aims Adult patients suffering from multimorbidity are at high risk of medication non-adherence. It has been well established that self-management support is an effective strategy to enhance medication adherence for patients with chronic conditions. However, little is known about the effect of the medication self-management intervention in Adult patients with multimorbidity. The aim of this study to evaluate the effectiveness of a nurse-led medication self-management intervention in improving medication adherence and health outcomes in adult patients with multimorbidity.

Methods This study is a single centre, single-blind, two-arm randomised controlled trial. Adult patients with multi-morbidity will be recruited from NCCCR Qatar. A total of 100 participants will be randomly allocated to receive standard care or standard care plus the medication self-management intervention. The intervention will be delivered by clinical nurse specialists. The 6-week intervention includes three face-to-face education sessions (2st week, 4rd week and 6th week) and two weekly (8th week and 10 week) follow-up phone calls. Participants in the control group continue to receive all respects of standard care offered by healthcare providers, including chronic disease management, drug prescription, referral to hospital specialists, health education and consultations regarding patients' diseases and treatments during centre visits.

Outcome The primary outcome is medication adherence as measured by the 8-item Medication Adherence Report Scale. Secondary outcomes include medication self-management capacity (medication knowledge, medication beliefs, and medication self-efficacy), treatment experiences (medication treatment satisfaction and treatment burden). All outcomes will be measured at baseline, immediately post-intervention (7th week), and at 3-month post-intervention.

DETAILED DESCRIPTION:
In terms of intervention we are giving six weeks motivational training ( 3 face face session and 2 telephonic follow ups).

ELIGIBILITY:
Inclusion Criteria:

* +18 years old or over,
* Patients with at least two of the identified comorbidities (Hypertension, Chronic painful condition, Cancer, Inflammatory connective tissue disorders, Diabetes, Lipid disorder, Dyspepsia and gastroenteritis, Heart disease, Chronic obstructive pulmonary disease, Stroke and cerebrovascular disease , chronic kidney disorder , Asthma Thyroid disorders, Anemia, Chronic liver disease, Depression, Epilepsy, Anxiety & other stress related disorders), (3) having at least one medication prescribed for a chronic condition over at least the 3 months prior to inclusion in the study,
* Non-adherence to medications, as defined by scoring zero on the 8-item Medication Adherence Report Scale (Morisky -8)(29),
* Independently managing their medications (i.e., not rely on a care taker),
* Able to speak or understand English/Arabic,
* Able and willing to receive phone calls, and
* Capable of providing a written informed consent to participate in the study.

Exclusion Criteria:

* Being institutionalized in a long-term care facility,
* Planning to move away from the community in the next 6 months,
* Cognitive impairment (Mini-cog scores < 4), and
* Currently participating in research involving chronic disease management. Patients with cognitive impairment are excluded because they may not be able to provide valid answers to the questionnaires.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Medication Adherence | 3 months
  The Morisky-8 is a self-reporting measure of unintentional and intentional medication non-adherent behaviors with a yes and no response. The total score of the moresky-8 ranges from 0 to 8, with a higher score representing higher adherence to medication. Approx 50% percentage change in medication adherence after intervention from baseline to 3 months as compared to control

SECONDARY OUTCOMES:
Medication Knowledge | 3 months
  Change medication knowledge using The Patients' Perceived Knowledge in Medication Use Questionnaire (PKMUQ). The response scale ranges from 1 = strongly disagree to 5 = strongly agree, and the response scores of all 5 items will be summed. Higher scores indicate a higher level of medication knowledge. the score will vary from 5 to 25.
Medication beliefs | 3 months
  using the Beliefs about Medication Questionnaire (BMQ 18-item)self-reported questionnaire we will assess the medication beliefs from baseline to 3 months.
  A 5-point Likert scale ranging from 1 = strongly disagree to 5 = strongly agree is used. A higher score indicates stronger beliefs about the corresponding concepts in each subscale. the score range would be 5 to 90.
Medication self-efficacy | 3 months
  Change in Self efficacy will be assess using the SEAMS 13 items of questionnaire. Each item has a 3-point scale ranging from 1 = not confident to 3 = very confident. The score of scale ranges from 13 to 39, with a higher medication self-efficacy by a higher score.
Treatment burden | 3 months
  The change in behavior and emotional burden using MTBQ questionnaire. Each item is scored on 6-point Likert scale, ranging from 0 = does not apply to 5 = most difficult. Scores are summed to derive a total score ranging from 0 to 50 with a higher score indicating a higher level of treatment burden.

IPD SHARING:
Plan to Share IPD: No
Research data will be stored on a password-protected computer and backed up on a password-protected hard drive Research Department 322A 3rd floor 302.
  PI and Senior Biostatistician will have the access of full data

REFERENCES:
- [Derived] Singh K, Joy GV, Al Bulushi A, Alomari AMA, Mannethodi K, Kunjavara J, Hassan N, Idris Z, Yassin MADM, Al Lenjawi B. Nurse-led medication self-management intervention in the improvement of medication adherence in adult patients with multi-morbidity: A Protocol for a Feasibility Randomized controlled trial. Glob Epidemiol. 2025 Jan 9;9:100184. doi: 10.1016/j.gloepi.2025.100184. eCollection 2025 Jun. PMID 39897388

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-02): https://cdn.clinicaltrials.gov/large-docs/53/NCT05645653/Prot_SAP_000.pdf
  • Informed Consent Form (2022-11-02): https://cdn.clinicaltrials.gov/large-docs/53/NCT05645653/ICF_001.pdf